CLINICAL TRIAL: NCT07203157
Title: A Pilot Study Evaluating the Effect and Feasibility of Virtual Reiki Therapy as a Complementary Treatment for Patients With Systemic Lupus Erythematosus
Brief Title: HEAL-SLE: Holistic Energy for Alleviating Lupus Symptoms
Acronym: HEAL-SLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Daisy Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-00357
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE; Reiki
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reiki Therapy (Experimental): Participants receiving standard of care (SOC) treatment for SLE will continue SOC while receiving research-specific Virtual Reiki therapy once per week for 8 weeks.
  Interventions: Other: Virtual Reiki Therapy

INTERVENTIONS:
Other: Virtual Reiki Therapy — 20-minute session once per week for 8 weeks via Webex. Each session will be delivered remotely by a Certified Reiki Practitioner Level II or higher.

SUMMARY:
The purpose of this study is to assess the efficacy, feasibility, and acceptability of Virtual Reiki therapy as a complementary treatment for patients with systemic lupus erythematosus (SLE). The study also aims to investigate the feasibility, acceptability, and adherence of integrating Virtual Reiki therapy within the healthcare system for patients with SLE. Participants receiving standard of care (SOC) treatment for SLE will continue SOC while receiving research-specific Virtual Reiki therapy once per week for 8 weeks. Each study session will be delivered remotely by a Certified Reiki Practitioner Level II or higher.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 and older at the time of informed consent
2. Diagnosed with SLE (based on 2019 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) criteria)
3. Currently receiving SOC treatment for SLE at NYU Langone Orthopedic Center
4. Able and willing to provide consent and participate in 8 weekly virtual Reiki sessions
5. Has access to reliable internet, have an active email address, and able to utilize WebEx
6. Able to read, speak and understand English

Exclusion Criteria:

1. Under 18 years of age
2. Patients experiencing severe disease activity requiring hospitalization at time of screening
3. Unable to read, speak and understand English
4. No access to internet
5. Not willing to participate in weekly virtual Reiki sessions
6. Currently enrolled in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scales (VAS) score | Baseline, Week 4
  VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Change in Visual Analog Scales (VAS) score | Week 4, Week 8
  VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 10 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.

SECONDARY OUTCOMES:
Number of Reiki sessions completed over the 8-week period | Week 8
  Adherence will be measured using a reiki visit log to monitor the number of Reiki sessions completed over the 8- week period. Participants completing fewer than 75% of scheduled sessions (fewer than 6 out of 8 sessions) will be excluded from the final analysis to ensure study data integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gamez-Perez, RN, BSN, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Monica.Gamez-Perez@NYULangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Monica.Gamez-Perez@NYULangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.